CLINICAL TRIAL: NCT01223183
Title: Absorptive Clearance After Inhaled Osmotics in Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tim Corcoran, PhD, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRO09080375
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; nuclear medicine; aerosol; nebulizer
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects inhale isotonic saline on one imaging day and 7% hypertonic on the other. The order is randomized. There is a period of 5-24 days between imaging days.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- isotonic saline then hypertonic saline (Active Comparator): Subjects inhaled nebulized isotonic saline on study day 1, and then after a 5-24 day washout period, subjects inhaled nebulized 7% hypertonic saline on study day 2.
  Interventions: Drug: hypertonic saline (7%); Drug: isotonic saline
- hypertonic saline then isotonic saline (Active Comparator): Subjects inhaled nebulized 7% hypertonic saline on study day 1, and then after a 5-24 day washout period, subjects inhaled nebulized isotonic saline on study day 2.
  Interventions: Drug: hypertonic saline (7%); Drug: isotonic saline

INTERVENTIONS:
Drug: hypertonic saline (7%) — single treatment by inhalation
Drug: isotonic saline — single treatment by inhalation

SUMMARY:
Blockage of the breathing tubes of the lungs by thick, sticky mucus is a major cause of lung problems for people with cystic fibrosis (CF). Many researchers now believe that people with CF absorb too much water from the insides of their lungs, and that the mucus in their lungs becomes so thick and sticky because there is not enough water in it. The investigators are trying to develop ways to measure how fast water is absorbed from the breathing tubes in the lung so that the investigators can more quickly test new medications that are being developed to fix this problem for CF patients. The investigators have already done studies showing that people with CF absorb a particular radioactive drug (Indium-111 diethylenetriaminepentaacetic acid or In-DTPA) from their lungs more quickly than people without CF. Now the investigators are trying to prove that the absorption of this drug is related to the absorption of water. The investigators measure the absorption of In-DTPA by delivering it in an aerosol (inhaled mist) along with another radioactive drug (Technetium 99m sulfur colloid or Tc-SC). This other drug helps us measure how much material is cleared from the lungs in other ways (like coughing) without being absorbed. In this study, the investigators will measure how the absorption of In-DTPA is affected by inhaling isotonic saline and hypertonic saline (salt water), both of which the investigators know affect the absorption of water in the airways.

DETAILED DESCRIPTION:
There is a substantial need for new biomarkers in the study of cystic fibrosis (CF) lung disease. Conventional endpoints, such as rate of FEV1 decline, require prolonged trials and large sample sizes to demonstrate therapeutic efficacy. Ideally such biomarkers would provide a quantitative window to the most basic aspects of CF pathophysiology, allowing for the development and evaluation of therapies prior to large scale clinical trials. The basic defect of CF lung disease occurs in the airways where dysfunction of the cystic fibrosis transmembrane conductance regulator (CFTR) and epithelial sodium (ENaC) channels is thought to create an ionic gradient that causes excessive liquid absorption across the epithelium. This results in a dehydrated airway surface liquid (ASL) layer, defective mucociliary clearance, and an increased proclivity for infection and inflammation.

Aerosol-based methods have been developed to measure mucociliary clearance in the lung and used to demonstrate the efficacy of inhaled osmotic therapies. We have developed an aerosol technique to measure both mucociliary clearance and the absorptive clearance of a hydrophilic small molecule (diethylenetriaminepentaacetic acid or DTPA) in whole, central, and peripheral lung regions. We estimate DTPA absorption by delivering an aerosol containing both Indium 111 DTPA (In-DTPA) and Technetium 99m sulfur colloid (Tc-SC) to the airways. The clearance of each radiopharmaceutical is imaged independently and two separate clearance curves are calculated. In-DTPA is cleared through both absorption and mucociliary clearance while Tc-SC is cleared only through the mucociliary route. The difference between the clearance rates of the radiopharmaceuticals provides an estimate of In-DTPA absorption rate.

Our previous studies have demonstrated that absorption of In-DTPA occurs at a higher rate in central (airway dominated) lung zones of CF subjects compared to controls (42 vs. 32 %/hr, CF n= 9, control n=10, p=0.03). We believe that this increased In-DTPA absorption is being caused by the increased liquid absorption occurring in these airways, however there are other potential causes such as increase in tight junction permeability or epithelial denuding.

In this study we propose to measure In-DTPA absorption after the delivery of interventions known to affect liquid absorption in the airways to see if changes in In-DTPA absorption mirror the changes in liquid absorption known to be caused by the interventions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms
* clinically stable as determined by the investigator (pulmonologist)

Exclusion Criteria:

* intolerant to hypertonic saline.
* FEV1%p <40% of predicted
* nursing mother
* positive urine pregnancy test
* unwilling to stop hypertonic saline therapy for 72 hours prior to each test day
* cigarette smoker (regular smoking within 6 months of study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Corcoran, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corcoran TE, Thomas KM, Myerburg MM, Muthukrishnan A, Weber L, Frizzell R, Pilewski JM. Absorptive clearance of DTPA as an aerosol-based biomarker in the cystic fibrosis airway. Eur Respir J. 2010 Apr;35(4):781-6. doi: 10.1183/09031936.00059009. Epub 2009 Aug 28. PMID 19717485
- [Result] Locke LW, Myerburg MM, Markovetz MR, Parker RS, Weber L, Czachowski MR, Harding TJ, Brown SL, Nero JA, Pilewski JM, Corcoran TE. Quantitative imaging of airway liquid absorption in cystic fibrosis. Eur Respir J. 2014 Sep;44(3):675-84. doi: 10.1183/09031936.00220513. Epub 2014 Apr 17. PMID 24743971
- [Derived] Locke LW, Myerburg MM, Weiner DJ, Markovetz MR, Parker RS, Muthukrishnan A, Weber L, Czachowski MR, Lacy RT, Pilewski JM, Corcoran TE. Pseudomonas infection and mucociliary and absorptive clearance in the cystic fibrosis lung. Eur Respir J. 2016 May;47(5):1392-401. doi: 10.1183/13993003.01880-2015. Epub 2016 Mar 23. PMID 27009167

RESULTS

PARTICIPANT FLOW:
Groups:
- Isotonic Saline Then Hypertonic Saline: Subjects inhale nebulized isotonic saline on study day 1, then perform a washout period of 5-24 days, then inhale 7% hypertonic saline on study day 2.
- Hypertonic Saline Then Isotonic Saline: Subjects inhale nebulized 7% hypertonic saline on study day 1, then perform a 5-24 day washout period, and then inhale nebulized isotonic saline on study day 2.
Period: Imaging Day 1
Arm/Group | Isotonic Saline Then Hypertonic Saline | Hypertonic Saline Then Isotonic Saline
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Washout Period (5-24 Days)
Arm/Group | Isotonic Saline Then Hypertonic Saline | Hypertonic Saline Then Isotonic Saline
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Imaging Day 2
Arm/Group | Isotonic Saline Then Hypertonic Saline | Hypertonic Saline Then Isotonic Saline
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Isotonic Saline Then Hypertonic Saline: Subjects inhaled isotonic saline on study day 1, then had a washout period of 5-24 days, then inhaled 7% hypertonic saline on study day 2
- Hypertonic Saline Then Isotonic Saline: Subjects inhaled 7% hypertonic saline on study day 1, then had a washout period of 5-24 days, then inhaled isotonic saline on study day 2
- Total: Total of all reporting groups
Arm/Group | Isotonic Saline Then Hypertonic Saline | Hypertonic Saline Then Isotonic Saline | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (11) | 24 (5) | 26 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Absorptive Clearance Rate After Isotonic Saline Inhalation
Description: The absorption rate of Indium 111 diethylenetriaminepentaacetic acid (In-DTPA) in the airways after the inhalation of isotonic saline
Time Frame: 80 minutes after radiopharmaceutical inhalation
Population: This group includes data from the isotonic saline inhalation day from both the "isotonic then hypertonic" and the "hypertonic than isotonic" groups who had sufficient imaging data to allow for full analysis.
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Groups:
- Isotonic Saline Inhalation: Results from isotonic inhalation day
Arm/Group | Isotonic Saline Inhalation
Number analyzed (Participants) | 12
percent cleared / 80 minutes | 32.0 (13.9)

2. Primary Outcome: Absorptive Clearance Rate After Hypertonic Saline Inhalation
Description: The absorption rate of In-DTPA after the inhalation of hypertonic saline
Time Frame: 80 minutes after radiopharmaceutical inhalation
Population: This group includes data from the hypertonic saline inhalation day from both the "isotonic then hypertonic" and the "hypertonic than isotonic" groups who had sufficient imaging data to allow for full analysis.
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Groups:
- Hypertonic Saline Inhalation: Results from hypertonic saline inhalation day
Arm/Group | Hypertonic Saline Inhalation
Number analyzed (Participants) | 11
percent cleared / 80 minutes | 22.2 (12.8)
Statistical Analysis 1: Comparison: Hypertonic Saline Inhalation; Comparing DTPA absorption after hypertonic saline inhalation to DTPA absorption after isotonic saline inhalation; Test type: Equivalence — alpha=0.05; p < 0.001, t-test, 2 sided

3. Primary Outcome: Mucociliary Clearance Rate After Isotonic Saline Inhalation
Description: The clearance rate of Tc-SC after the inhalation of isotonic saline
Time Frame: 80 minutes after radiopharmaceutical inhalation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Groups:
- Isotonic Saline Inhalation: Results from isotonic saline inhalation day
Arm/Group | Isotonic Saline Inhalation
Number analyzed (Participants) | 12
percent cleared / 80 minutes | 23.6 (10.3)

4. Primary Outcome: Mucociliary Clearance Rate After Hypertonic Saline Inhalation
Description: The clearance rate of Tc-SC after the inhalation of hypertonic saline
Time Frame: 80 minutes after radiopharmaceutical inhalation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Arm/Group | Hypertonic Saline Inhalation
Number analyzed (Participants) | 11
percent cleared / 80 minutes | 42.4 (18.2)
Statistical Analysis 1: Comparison: Hypertonic Saline Inhalation; Comparing mucociliary clearance after isotonic saline inhalation to mucociliary clearance after hypertonic saline inhalation; Test type: Equivalence — alpha=0.05; p = 0.003, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the start of imaging day 1 to the end of imaging day 2
Groups:
- Isotonic Saline Then Hypertonic Saline: Subjects inhaled isotonic saline on study day 1 and hypertonic saline on study day 2
- Hypertonic Saline Then Isotonic Saline: Subjects inhaled hypertonic saline on study day 1 and isotonic saline on study day 2
Arm/Group | Isotonic Saline Then Hypertonic Saline | Hypertonic Saline Then Isotonic Saline
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isotonic Saline Then Hypertonic Saline (N=10) | Hypertonic Saline Then Isotonic Saline (N=10)
hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalization unrelated to study procedures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isotonic Saline Then Hypertonic Saline (N=10) | Hypertonic Saline Then Isotonic Saline (N=10)
hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Subject was hospitalized between imaging days due to a problem not related to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes